CLINICAL TRIAL: NCT03372057
Title: A Multi-Center, Phase 2, Open-label, Parallel Cohort Study of Efficacy and Safety of Duvelisib in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma (PTCL)
Brief Title: A Study of Duvelisib in Participants With Relapsed or Refractory Peripheral T-cell Lymphoma (PTCL)
Acronym: PRIMO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VS-0145-225; 2019-001123-13 (EudraCT Number)
Record Dates: First submitted 2017-12-01; First posted 2017-12-13 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: Lymphoma; T-cell Lymphoma; Relapse; Refractory; PI3K-δ,γ
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma; Lymphoma, T-Cell; Recurrence | interventions — duvelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Optimization Phase: Cohort 1 (Experimental): Duvelisib PO BID at a starting dose of 25 mg, with potential escalation on a per-participant basis to 50 mg and then 75 mg, based on the participant's response to and tolerance of therapy, in 28-day cycles.
  Interventions: Drug: Duvelisib
- Dose Optimization Phase: Cohort 2 (Experimental): Duvelisib 75 mg PO BID, administered in 28-day cycles.
  Interventions: Drug: Duvelisib
- Expansion Phase (Experimental): Duvelisib PO BID at a starting dose of 75 mg for the first 2 cycles, followed by a mandatory reduction to 25 mg BID thereafter for those participants with complete response (CR), partial response (PR) or stable disease (SD), in 28-day cycles (dose determined in Optimization Phase).
  Interventions: Drug: Duvelisib

INTERVENTIONS:
Drug: Duvelisib — Duvelisib PO 25 mg BID or 50 mg BID or 75 mg BID in 28-day cycles.
  Other Names: IPI-145
  Arms: Dose Optimization Phase: Cohort 1
Drug: Duvelisib — Duvelisib PO 75 mg BID in 28-day cycles.
  Other Names: IPI-145
  Arms: Dose Optimization Phase: Cohort 2
Drug: Duvelisib — Duvelisib PO BID in 28-day cycles (dose determined in Optimization Phase).
  Other Names: IPI-145
  Arms: Expansion Phase

SUMMARY:
This is a multi-center, parallel cohort, open-label, Phase 2 study of duvelisib, an oral dual inhibitor of phosphoinositide-3-kinase-delta, gamma (PI3K-δ,γ), in participants with relapsed/refractory peripheral T-cell lymphoma (PTCL).

DETAILED DESCRIPTION:
The study had 2 phases, a Dose Optimization Phase and an Expansion Phase.

In the Dose Optimization Phase, participants were randomly assigned to 1 of 2 study cohorts, as follows:

* Cohort 1: Duvelisib per oral (PO) twice daily (BID) at a starting dose of 25 milligrams (mg), with potential escalation on a per-participant basis to 50 mg and then 75 mg, based on the participant's response to and tolerance of therapy, in 28-day cycles.
* Cohort 2: Duvelisib 75 mg PO BID, administered in 28-day cycles.

A total of 20 participants were to be enrolled in the Dose Optimization Phase, with 10 participants per cohort. Based on the safety and activity data obtained in the Dose Optimization Phase of the study, the Expansion Phase dose of duvelisib was to be determined.

In the Expansion Phase, approximately 100-130 participants were to be enrolled and receive duvelisib dose in 28-day cycles as determined in Dose Optimization Phase.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age
2. Diagnosis of one of the following histologic subtypes of PTCL, pathologically confirmed, as defined by the World Health Organization:

   1. Peripheral T-cell lymphoma-not otherwise specified;
   2. Angioimmunoblastic T-cell lymphomas;
   3. Anaplastic large cell lymphoma (ALCL); or
   4. Natural-killer/T-cell lymphoma
3. Received at least 2 cycles of one standard regimen for newly diagnosed advanced PTCL, and one of the following:

   1. failed to achieve at least a PR after 2 or more cycles of standard therapy;
   2. failed to achieve a CR after completion of standard therapy; and/or
   3. persistent or progressive disease after an initial response
4. For participants with CD30+ ALCL, failed or are ineligible or intolerant to brentuximab vedotin
5. Measurable disease as defined by Lugano for PTCL, that is, at least 1 measurable disease lesion > 1.5 centimeters in at least one dimension by conventional techniques (fluorine-18 fluorodeoxyglucose positron emission tomography/computed tomography [CT], CT with contrast, magnetic imaging resonance)

Exclusion Criteria:

1. Primary leukemic PTCL subtypes (that is, T-cell prolymphocytic leukemia, T-cell large granular lymphocytic leukemia, adult T-cell leukemia/lymphoma and aggressive NK-cell leukemia) or transformed mycosis fungoides
2. Received prior allogeneic transplant
3. Received prior treatment with a PI3K inhibitor
4. Known central nervous system involvement by PTCL
5. Ongoing treatment with chronic immunosuppressants (e.g., cyclosporine) or systemic steroids > 20 mg of prednisone (or equivalent) once daily
6. Ongoing treatment for systemic bacterial, fungal, or viral infection at Screening
7. Known hypersensitivity to duvelisib and/or its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (19):
  - City of Hope National Medical Center, Duarte, California
  - University of California - Irvine, Irvine, California
  - University of California - Los Angeles, Los Angeles, California
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University - Feinberg School of Medicine, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - The Ohio State University, Columbia, Ohio
  - Toledo Cancer Center, Toledo, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Baylor Research Institute - Charles Sammons Cancer Center, Dallas, Texas
- Germany (2):
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Universitätsklinikum Halle (Saale) - Klinik und Poliklinik für Innere Medizin IV, Halle, Saxony-Anhalt
- Italy (5):
  - ASST Papa Giovanni XXIII - Medicina Trasfusionale ed Ematologia - Bergamo, Bergamo
  - A.O.di Bologna Policl.S.Orsola, Bologna
  - Ieo, Irccs, Milan
  - Policlinico Universitario Agostino Gemelli, Università Cattolica del Sacro Cuore, Roma
  - Azienda Ospedaliera Santa Maria di Terni, Terni
- Japan (8):
  - Japanese Site 8, Fukuoka
  - Japanese Site 5, Kobe
  - Japanese Site 3, Miyagi
  - Japanese Site 6, Nagoya
  - Japanese Site 7, Niigata
  - Japanese Site 1, Okayama
  - Japanese Site 2, Tokyo
  - Japanese Site 4, Tokyo
- United Kingdom (2):
  - Christie Hospital NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Regardless of study phase, all participants underwent screening assessments up to 30 days before the first study drug dose.
Groups:
- Dose Optimization Phase: Cohort 1: Duvelisib was administered orally (PO) twice daily (BID) at a starting dose of 25 milligrams (mg), with potential escalation on a per-participant basis to 50 mg and then 75 mg, based on the participant's response to and tolerance of therapy, in 28-day cycles.
- Dose Optimization Phase: Cohort 2: Duvelisib 75 mg PO BID was administered in 28-day cycles.
- Expansion Phase: Duvelisib PO BID at a starting dose of 75 mg was administered for the first 2 cycles (28-day cycles), followed by a mandatory reduction to 25 mg BID thereafter for those participants with complete response (CR), partial response (PR) or stable disease (SD), in 28-day cycles (dose determined in Optimization Phase).
Period: Dose Optimization Phase
Arm/Group | Dose Optimization Phase: Cohort 1 | Dose Optimization Phase: Cohort 2 | Expansion Phase
Started | 20 | 13 | 0
Received at Least 1 Dose of Study Drug (Safety Analysis Set; Modified Intent-to-treat (mITT)) | 20 | 13 | 0
Completed | 0 | 0 | 0
Not Completed | 20 | 13 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Closure Of The Study By The Sponsor | 3 | 1 | 0
Not completed — Death | 16 | 11 | 0
Period: Expansion Phase
Arm/Group | Dose Optimization Phase: Cohort 1 | Dose Optimization Phase: Cohort 2 | Expansion Phase
Started | 0 | 0 | 123 (Participants enrolled for Expansion Phase only.)
Received at Least 1 Dose of Study Drug (Safety Analysis Set; Modified Intent-to-treat (mITT)) | 0 | 0 | 123
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 123
Not completed — Withdrawal by Subject | 0 | 0 | 4
Not completed — Closure Of The Study By The Sponsor | 0 | 0 | 39
Not completed — Death | 0 | 0 | 78
Not completed — Progressive Disease | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who received at least one dose of study drug.
Groups:
- Expansion Phase: Duvelisib PO BID at a starting dose of 75 mg for the first 2 cycles, followed by a mandatory reduction to 25 mg BID thereafter for those participants with CR, PR or SD, in 28-day cycles (dose determined in Optimization Phase).
- Total: Total of all reporting groups
Arm/Group | Dose Optimization Phase: Cohort 1 | Dose Optimization Phase: Cohort 2 | Expansion Phase | Total
Number analyzed (Participants) | 20 | 13 | 123 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (14.81) | 65.0 (7.22) | 62.9 (13.59) | 63.2 (13.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 56 | 66
  Male | 14 | 9 | 67 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 12 | 14
  Not Hispanic or Latino | 18 | 12 | 111 | 141
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 18 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 9 | 11
  White | 16 | 12 | 92 | 120
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 4 | 5
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG Performance Status: a scale that measures how cancer affects a participant's daily living abilities. The scale ranges from 0 (fully active) to 5 (dead). 0 = fully active without restriction; 1 = Restricted in physically strenuous activity; 2 = Ambulatory, capable of all selfcare; 3 = Capable of limited selfcare; 4 = Completely disabled; 5 = Dead.
  participants
    0 | 8 | 5 | 49 | 62
    1 | 8 | 7 | 64 | 79
    2 | 3 | 1 | 10 | 14
    3 | 0 | 0 | 0 | 0
    4 | 0 | 0 | 0 | 0
    5 | 0 | 0 | 0 | 0
    Missing | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) as Assessed by the Investigator Using the Lugano Criteria
Description: ORR was defined as the percentage of participants with CR + PR, as assessed by the investigator using the Lugano criteria, for participants receiving the optimal dose of duvelisib for at least one cycle of study therapy.
Time Frame: 56 days (2 cycles; 28-day cycles)
Population: Dose Optimization Efficacy Set: All participants who received at least one dose of study drug, completed at least one cycle of treatment, and had at least one scan to assess disease response after completion of one cycle of treatment. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure. As pre-specified, efficacy analysis using investigator assessment reported for the Dose Optimization Phase only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Optimization Phase: Cohort 1 | Dose Optimization Phase: Cohort 2
Number analyzed (Participants) | 13 | 13
percentage of participants | 53.8 [26.7 to 80.9] | 53.8 [26.7 to 80.9]

2. Primary Outcome: ORR as Assessed by the Independent Review Committee (IRC) Using the Lugano Criteria
Description: ORR was defined as the percentage of participants with CR + PR, as assessed by the IRC using the Lugano criteria, for participants receiving the optimal dose of duvelisib for at least one cycle of study therapy.
Time Frame: 56 days (2 cycles; 28-day cycles)
Population: Modified Intent-to-treat (mITT): all participants who received at least one dose of study drug. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure. As pre-specified, efficacy analysis using IRC assessment reported for the Expansion Phase only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Expansion Phase
Number analyzed (Participants) | 123
percentage of participants | 48.0 [39.1 to 56.8]

3. Secondary Outcome: Duration of Response (DOR) as Assessed by the Investigator Using the Lugano Criteria
Description: DOR was defined for participants with CR or PR as the time from the date of the first documentation of response (CR or PR) to the date of the first documentation of progressive disease (PD) or death due to any cause. Participants who withdraw from the study for any reason prior to PD and participants who had ongoing response at the time of the data cut were censored at the date of their last response assessment.
Time Frame: Up to 70 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Dose Optimization Phase: Cohort 1 | Dose Optimization Phase: Cohort 2
Number analyzed (Participants) | 5 | 5
month | 4.22 [1.87 to NA] — Insufficient number of participants with events to calculate upper confidence intervals. | 3.32 [1.77 to NA] — Insufficient number of participants with events to calculate upper confidence intervals.

4. Secondary Outcome: Progression-free Survival (PFS) as Assessed by the Investigator Using the Lugano Criteria
Description: PFS was defined as the time from the date of first treatment to the date of the first radiographic disease progression or death due to any cause, whichever occurred first.
Time Frame: Up to 70 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Dose Optimization Phase: Cohort 1 | Dose Optimization Phase: Cohort 2
Number analyzed (Participants) | 10 | 11
month | 3.55 [1.05 to 8.54] | 3.55 [1.81 to 13.14]

5. Secondary Outcome: Disease Control Rate (DCR) As Assessed by the Investigator Using the Lugano Criteria
Description: DCR was defined as the percentage of participants with a best overall response of CR or PR or with a best overall response of stable disease (SD) sustained for at least 8 weeks.
Time Frame: Up to 8 weeks
Population: Dose Optimization Efficacy Set: All participants who received at least one dose of study drug, completed at least one cycle of treatment, and had at least one scan to assess disease response after completion of one cycle of treatment. As pre-specified, efficacy analysis using investigator assessment reported for the Dose Optimization Phase only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Optimization Phase: Cohort 1 | Dose Optimization Phase: Cohort 2
Number analyzed (Participants) | 13 | 13
percentage of participants | 61.5 [35.1 to 88.0] | 61.5 [35.1 to 88.0]

6. Secondary Outcome: DOR as Assessed by the IRC Using the Lugano Criteria
Description: DOR was defined for participants with CR or PR as the time from the date of the first documentation of response (CR or PR) to the date of the first documentation of PD or death due to any cause. Participants who withdrew from the study for any reason prior to PD and participants who had ongoing response at the time of the data cut were censored at the date of their last response assessment.
Time Frame: Up to 70 months
Population: Modified Intent-to-treat (mITT): all participants who receive at least one dose of study drug. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure. As pre-specified, efficacy analysis using IRC assessment reported for the Expansion Phase only.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Expansion Phase
Number analyzed (Participants) | 25
month | 7.9 [6.4 to 21.00]

7. Secondary Outcome: PFS as Assessed by the IRC Using the Lugano Criteria
Description: as for outcome 4
Time Frame: Up to 70 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Expansion Phase
Number analyzed (Participants) | 74
months | 3.4 [1.8 to 3.9]

8. Secondary Outcome: DCR as Assessed by the IRC Using the Lugano Criteria
Description: DCR was defined as the percentage of participants with a best overall response of CR or PR or with a best overall response of SD sustained for at least 8 weeks.
Time Frame: Up to 8 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Expansion Phase
Number analyzed (Participants) | 123
percentage of participants | 49.6 [40.8 to 58.4]

9. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first treatment to the date of death due to any cause. Participants without documented death were censored at last alive date.
Time Frame: Up to 70 months
Population: Dose Optimization Efficacy Set: All participants who received at least one dose of study drug, completed at least one cycle of treatment, and had at least one scan to assess disease response after completion of one cycle of treatment. Modified Intent-to-treat (mITT): all participants who receive at least one dose of study drug. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Dose Optimization Phase: Cohort 1 | Dose Optimization Phase: Cohort 2 | Expansion Phase
Number analyzed (Participants) | 9 | 11 | 78
month | 6.70 [5.22 to NA] — Insufficient number of participants with events to calculate the upper confidence interval. | 10.58 [6.67 to 44.62] | 12.4 [8.4 to 22.7]

10. Secondary Outcome: Plasma Concentration of IPI-145 (Duvelisib) and IPI-656 (Metabolite)
Description: Blood samples were taken for the analyses of duvelisib and IPI-656 in plasma at designated time points. Results are reported as nanograms/milliliter (ng/mL).
Time Frame: Day 15 of Cycles 1 and 2 (4 hours postdose) (28-day cycles)
Population: Safety Analysis Set: all participants who received at least one dose of study drug. Here, 'Overall Number of Participants Analyzed' signifies those who were evaluable for this outcome measure, and 'Number Analyzed' signifies those participants who were evaluable for this outcome measure at the specified time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Optimization Phase: Cohort 1 | Dose Optimization Phase: Cohort 2 | Expansion Phase
Number analyzed (Participants) | 14 | 12 | 100
ng/mL
  Duvelisib: Cycle 1, Day 15 | 1238.1 (787.53) | 2070.0 (889.39) | 2873.7 (1709.15)
  Duvelisib: Cycle 2, Day 15: number analyzed (Participants) | 4 | 0 | 68
  Duvelisib: Cycle 2, Day 15 | 1492.5 (1019.10) |  | 2648.2 (1336.94)
  Metabolite (IPI-156): Cycle 1, Day 15 | 1310.4 (1408.99) | 1580.9 (772.13) | 2387.5 (1919.33)
  Metabolite (IPI-156): Cycle 2, Day 15: number analyzed (Participants) | 4 | 0 | 68
  Metabolite (IPI-156): Cycle 2, Day 15 | 894.8 (441.55) |  | 2427.0 (1655.89)

ADVERSE EVENTS:
Time Frame: From start of treatment (Day 1) to end of study (70 months)
Description: All reported safety data based upon Safety Analysis Set: all participants who received at least one dose of study drug. All-cause mortality reported as occurrence of death due to any cause during the study and after study discontinuation.
Arm/Group | Dose Optimization Phase: Cohort 1 | Dose Optimization Phase: Cohort 2 | Expansion Phase
All-Cause Mortality (participants affected / at risk) | 16/20 | 11/13 | 78/123
Serious Adverse Events (participants affected / at risk) | 14/20 | 9/13 | 60/123
Other Adverse Events (participants affected / at risk) | 19/20 | 13/13 | 121/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Optimization Phase: Cohort 1 (N=20) | Dose Optimization Phase: Cohort 2 (N=13) | Expansion Phase (N=123)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 9
Colitis (Gastrointestinal disorders) | 1 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Disease progression (General disorders) | 3 | 0 | 10
Pyrexia (General disorders) | 1 | 3 | 6
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 1
Chills (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 4 | 0 | 4
Sepsis (Infections and infestations) | 3 | 1 | 3
Bacteraemia (Infections and infestations) | 0 | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
COVID-19 (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Coronavirus infection (Infections and infestations) | 1 | 0 | 0
Cryptococcosis (Infections and infestations) | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1
Febrile infection (Infections and infestations) | 0 | 0 | 1
Herpes simplex viraemia (Infections and infestations) | 0 | 0 | 1
Infective spondylitis (Infections and infestations) | 0 | 0 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1
Systemic candida (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 3
Alanine aminotransferase increased (Investigations) | 1 | 0 | 3
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Epstein-Barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Vascular dementia (Nervous system disorders) | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Allogenic stem cell transplantation (Surgical and medical procedures) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Optimization Phase: Cohort 1 (N=20) | Dose Optimization Phase: Cohort 2 (N=13) | Expansion Phase (N=123)
Anaemia (Blood and lymphatic system disorders) | 7 | 5 | 34
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 7
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 2 | 7
Tachycardia (Cardiac disorders) | 1 | 2 | 4
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 2
Cataract (Eye disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 1 | 5
Eye irritation (Eye disorders) | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 4 | 13
Colitis (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 5 | 2 | 22
Diarrhoea (Gastrointestinal disorders) | 9 | 9 | 41
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 8
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 9
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 5
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 9 | 6 | 31
Oral pain (Gastrointestinal disorders) | 0 | 2 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 3 | 15
Vomiting (Gastrointestinal disorders) | 6 | 2 | 16
Chills (General disorders) | 2 | 1 | 8
Face oedema (General disorders) | 4 | 1 | 1
Fatigue (General disorders) | 7 | 6 | 38
Generalised oedema (General disorders) | 2 | 0 | 1
Malaise (General disorders) | 2 | 0 | 3
Oedema peripheral (General disorders) | 6 | 3 | 19
Pyrexia (General disorders) | 6 | 6 | 28
Swelling face (General disorders) | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 1 | 0
Hypogammaglobulinaemia (Immune system disorders) | 1 | 1 | 0
Adenovirus infection (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 7
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 2 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 1 | 2
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 2 | 2
Pneumonia (Infections and infestations) | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 5
Urinary tract infection (Infections and infestations) | 1 | 1 | 5
Alanine aminotransferase increased (Investigations) | 4 | 7 | 47
Amylase increased (Investigations) | 2 | 0 | 9
Aspartate aminotransferase increased (Investigations) | 4 | 5 | 45
Blood alkaline phosphatase increased (Investigations) | 4 | 1 | 12
Blood bilirubin increased (Investigations) | 1 | 1 | 10
Blood creatinine increased (Investigations) | 3 | 0 | 16
Blood culture positive (Investigations) | 0 | 1 | 1
Blood immunoglobulin G decreased (Investigations) | 0 | 1 | 0
Blood lactate dehydrogenase (Investigations) | 0 | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 2 | 1 | 20
Immunoglobulins decreased (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 3 | 0 | 13
Lymphocyte count decreased (Investigations) | 4 | 2 | 17
Neutrophil count decreased (Investigations) | 8 | 3 | 41
Platelet count decreased (Investigations) | 11 | 6 | 34
Urine output decreased (Investigations) | 2 | 0 | 0
Weight decreased (Investigations) | 3 | 3 | 8
Weight increased (Investigations) | 2 | 0 | 4
White blood cell count decreased (Investigations) | 7 | 3 | 25
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 11
Dehydration (Metabolism and nutrition disorders) | 1 | 4 | 4
Glucose tolerance impaired (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 12
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 1 | 7
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 3 | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 1 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 4 | 13
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2 | 15
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 2 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 9
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 5
Dizziness (Nervous system disorders) | 3 | 2 | 9
Dysgeusia (Nervous system disorders) | 2 | 1 | 10
Headache (Nervous system disorders) | 0 | 3 | 8
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 9
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 8
Presyncope (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 2 | 5
Confusional state (Psychiatric disorders) | 2 | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 0 | 10
Acute kidney injury (Renal and urinary disorders) | 3 | 1 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 17
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 11
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 3 | 13
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 4
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3 | 20
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 14
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 4 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 2 | 21
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
Hypertension (Vascular disorders) | 1 | 1 | 16
Hypotension (Vascular disorders) | 3 | 2 | 12
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT03372057/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT03372057/SAP_001.pdf